CLINICAL TRIAL: NCT06784973
Title: A Phase 2, Randomized, Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Obeldesivir in Participants From Birth to < 5 Years of Age With Respiratory Syncytial Virus (RSV) Infection
Brief Title: Study of Obeldesivir to Treat Children With Respiratory Syncytial Virus (RSV) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by Sponsor; the decision was not due to any safety findings.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-685-6883; 2024-517998-24 (Other: European Medicines Agency)
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obeldesivir (Experimental): Participants will receive an age and weight appropriate ODV dose based on their cohort/group assignment.
  Interventions: Drug: Obeldesivir
- Obeldesivir Placebo (Experimental): Participants will receive an age and weight appropriate ODV placebo dose based on their cohort/group assignment.
  Interventions: Drug: Obeldesivir Placebo

INTERVENTIONS:
Drug: Obeldesivir — Administered orally
  Other Names: ODV; GS-5245
  Arms: Obeldesivir
Drug: Obeldesivir Placebo — Administered orally
  Arms: Obeldesivir Placebo

SUMMARY:
The goal of this clinical study is to check if obeldesivir (ODV; GS-5245) is safe and well-tolerated by children with respiratory syncytial virus (RSV) infection. It will also look at how well ODV helps reduce the time it takes for children to feel better and for their RSV symptoms to improve.

The primary objectives of this study are: a) to evaluate the safety and tolerability of ODV in pediatric participants with RSV infection; b) To evaluate the efficacy of ODV on time to alleviation of targeted RSV symptoms in pediatric participants with RSV infection.

DETAILED DESCRIPTION:
Pediatric participants will be enrolled as follows:

* Cohort 1: Infants and children from 4 weeks postnatal age, weighing ≥ 1.5 kg to < 40 kg
* Cohort 2: Neonates, either born at term or preterm, weighing ≥ 1.5 kg to < 6 kg

ELIGIBILITY:
Key Inclusion Criteria:

* Participants assigned male or female at birth, from birth to < 5 years of age who meet one of the following criteria, where permitted according to local law and approved nationally and by relevant institutional review board or independent ethics committee:

  * Cohort 1: Infants and children from 4 weeks postnatal age, weighing ≥ 1.5 kg to < 40 kg
  * Cohort 2: Neonates, either born at term or preterm, weighing ≥ 1.5 kg to < 6 kg
* RSV infection diagnosis ≤ 3 days prior to randomization.
* Negative test for influenza A/B, and SARS-CoV-2 infection ≤ 7 days prior to randomization.
* Onset of RSV signs or symptoms ≤ 3 days prior to randomization.
* Presence of at least 1 sign or symptom of RSV infection at screening and at randomization.

Key Exclusion Criteria:

* Currently requiring or expected to require hospitalization for RSV infection within 48 hours after randomization.
* Documented previous infection and/or hospitalization for RSV during the current respiratory virus season.
* Diagnosed with acute concurrent active systemic infections requiring treatment with systemic antiviral, antibacterial, antifungal, or antimycobacterial therapy, or with any documented respiratory viral infection (other than RSV), ≤ 7 days prior to randomization.
* History of asthma or recurrent wheezing.
* Neuromuscular disease that affects swallowing.
* Cystic fibrosis.
* Participants who are immunocompromised.
* Alanine aminotransferase ≥ 5 × upper limit of normal (ULN).
* Abnormal renal function.
* Concurrent or previous treatment with other agents with actual or possible direct antiviral activity against RSV, received within 28 days or within 5 half-lives, whichever is longer, prior to randomization.
* Received palivizumab within 100 days, or nirsevimab within 1 year, or other RSV specific monoclonal antibody within 5 half-lives of the antibody, prior to randomization.
* Participant whose mother received RSV vaccination during pregnancy and who is < 1 year old prior to randomization.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) Through Day 28 | First dose up to 28 days
Percentage of Participants Experiencing Grade 3 or 4 Treatment-emergent laboratory abnormalities by Day 28 | First dose up to 28 days
Time to Alleviation of Targeted RSV Symptoms by Day 28 | First dose up to 28 days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter AUCtau of ODV metabolite, GS-441524 | Day 1 to Day 5
  AUCtau is defined as the area under the concentration versus time curve over the dosing interval.
PK parameter Cmax of ODV metabolite, GS-441524 | Day 1 to Day 5
  Cmax is defined as the concentration at the end of the dosing interval.
PK parameter Ctrough of ODV metabolite, GS-441524 | Day 1 to Day 5
  Ctrough is defined as the concentration at the endo of the dosing interval.
Change From Baseline in RSV Nasal Swab Viral Load at Day 5 | Baseline, Day 5
Time to Sustained Alleviation of Targeted RSV Symptoms by Day 28 | First dose up to 28 days
Time to Resolution of Targeted RSV Symptoms by Day 28 | First dose up to 28days
Assessment of Palatability and Acceptability Scores of Age-specific Formulation as Assessed by Caregiver at Days 1 and 5 | Day 1 to Day 5
  Palatability and acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability and acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (55):
- United States (40):
  - Children's of Alabama, Birmingham, Alabama
  - Midway Medical Clinic, Oneonta, Alabama
  - Cohen Children's Medical Center Pharmacy New Pavillion, Phoenix, Arizona
  - Velocity Clinical Research, Phoenix, Phoenix, Arizona
  - UCLA (Outpatient Clinic), Los Angeles, California
  - Alliance Research Institute, Lynwood, California
  - Paradigm Clinical Research, Modesto, California
  - Paradigm Clinical Research Centers, LLC, San Diego, California
  - FOMAT - Jeffrey Kaplan MD Inc Pediatric Medicine, Santa Maria, California
  - Velocity Clinical Research, Washington DC, Washington D.C., District of Columbia
  - Dolphin Medical Research, Doral, Florida
  - Nona Pediatric Center, Orlando, Florida
  - PAS Research, Tampa, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - Velocity Clinical Research, Lafayette, Lafayette, Louisiana
  - Boeson Research, Great Falls, Montana
  - Boeson Research, Kalispell, Montana
  - Boeson Research, Missoula, Montana
  - Velocity Clinical Research - Norfolk, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Child Health Care Associates, Syracuse, New York
  - Epic Medical Research -Oklahoma, Chickasha, Oklahoma
  - Tekton Research, LLC, Yukon, Oklahoma
  - PAS Research, Pittsburgh, Pennsylvania
  - Helios Clinical Research, Burleson, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - PAS Research, Edinburg, Texas
  - Helios Clinical Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Sunrise Pediatrics, Houston, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - Pediatric Center, Richmond, Texas
  - Central Texas Medical Research, LLC, San Antonio, Texas
  - North Houston Internal Medicine and Pediatric Clinic, Tomball, Texas
  - Tanner Clinic, Kaysville, Utah
  - Tanner Clinic, Layton, Utah
  - Boeson Research PVU, Provo, Utah
- Japan (15):
  - Yoshimura Child Clinic, Akashi
  - Japan Community Healthcare Organization Kyushu Hospital, Fkitakyushu
  - Uchida child clinic, Fukuoka
  - Shindo Children's Clinic, Fukuoka
  - SEKI Children's CLINIC, Fukuoka
  - Ryuseidai Children's Clinic, Ibaraki
  - Isesaki Municipal Hospital, Isesaki
  - Abe Child Clinic, Kanagawa
  - Okada Kodomonomori Clinic, Kasukabe
  - Yutaka Children Clinic, Kobe
  - Kochi Health Sciences Center, Kochi
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya
  - Shimamura Memorial Hospital, Nerima-ku
  - Shizuoka Welfare Hospital, Shizuoka
  - Shizuoka City Shimizu Hospital, Shizuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06784973